CLINICAL TRIAL: NCT03169205
Title: Diabetes Mellitus With Pregnancy in Benisuef Localities
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Momen Zakaria Mohammed mohammed, assisstant lecturer, Beni-Suef University
Other Study IDs: 2500
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Pregnancy in Diabetics
MeSH Terms: conditions — Pregnancy in Diabetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- preexisting Diabetes mellitus type 1
  Interventions: Other: observation registry
- preexisting Diabetes mellitus type 2
  Interventions: Other: observation registry
- Gestational Diabetes mellitus
  Interventions: Other: observation registry

INTERVENTIONS:
Other: observation registry — observation registry

SUMMARY:
The aim of this work is to demonstrate the variation of Diabetes mellitus either preexisting or gestational Diabetes mellitus among pregnant ladies in our localities, detect maternal & fetal complications and to predict the risk factors for poor maternal, fetal & neonatal outcomes

ELIGIBILITY:
Inclusion Criteria:

* all pregnant ladies with Diabetes mellitus either type 1 or type 2
* all pregnant ladies with glucose intolerance which is first diagnosed during current pregnancy

Exclusion Criteria:

* ladies age less than 18 year or above 45

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: All pregnant ladies with impaired glucose intolerance either known before or fisrt diagnosed during current pregnancy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Maternal outcome | 2 years
  No. of patients who have preeclampsia,eclampsia,preterm delivery,Cesarean section,vaginal candidiasis,premature rupture of membrane,polyhydramnios,oligohydramnios,accidental hemorrhage,birth canal injuries,puerperal sepsis,wound infection,postpartum glucose intolerance.

SECONDARY OUTCOMES:
fetal outcome | 2 years
  No. of abortion,prematurity,macrosomia,congenital anomalies,intrauterine fetal death,still birth,shoulder dystocia,brachial plexus injury,neonatal death,respiratory distress syndrome,neonatal jaundice requiring photo-therapy,neonatal hypoglycemia,

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Banī Suwayf
  - Banī Suwayf